CLINICAL TRIAL: NCT04417426
Title: Sexual Behavior: Challenges in Prevention and Control Among Medical Students in Mexico
Brief Title: Sexual Behavior Among Medical Students in Mexico
Status: Completed | Type: Observational
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, GONZALEZ-OJEDA ALEJANDRO, Investigador Titular D, Instituto Mexicano del Seguro Social
Other Study IDs: STD01
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Sexually Transmitted Diseases
Keywords: Sexually transmitted diseases; Mass screening; Public health; Confounding Factors; Sexual intercourse; Epidemiologic
MeSH Terms: conditions — Sexually Transmitted Diseases; Coitus | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — A survey was conducted, which was filled voluntarily and completely anonymously; the demographic data asked were: sex, age, religion, and semester. We included questions about their sexual behavior: if they considered having enough knowledge about STDs, sexual intercourse onset, number of sexual partners in the last year, the total number of sexual partners, sexual orientation, the use of condoms and contraceptives, exclusive or non-exclusive sexual intercourses, frequency of STDs screening, and then if they know the location of STD testing centers.

SUMMARY:
This study aims to identify factors that influence students to undertake or not sexually transmitted diseases screening tests and to have an actual outlook of how Mexican university students live their sexual life. Moreover, the investigators aim to identify potential epidemiological risks and challenges to achieve adequate prevention and control of sexually transmitted diseases in this population. This is a descriptive cross-sectional study conducted at a private university in Guadalajara, Jalisco, Mexico, from December 2019 to April 2020.

DETAILED DESCRIPTION:
The investigators will invite the students to complete it and leave it in a black painted box to maintain privacy. The investigators will inquire if the participants considered having adequate knowledge about STDs, sexual intercourse onset, sexual behavior, number of sex partners, sexual orientation, use of condoms and contraceptives, sexual intercourse under the influence of alcohol or drugs, and reasons why students do not get sexually transmitted diseases screenings.

ELIGIBILITY:
Inclusion Criteria:

* University students currently attending medical school from 1st through 6th semester

Exclusion Criteria:

* Young adults not attending medical school
* Students out of the 1st - 6th-semester range

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Medical students attending a private university in Mexico from 1st through 6th semester
Sampling Method: Non-Probability Sample
Enrollment: 519 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-22 (Actual)

PRIMARY OUTCOMES:
Sexual intercourse onset | up to 4 months
  Age of first sexual relationship
Sexual partners in the last year | up to 4 months
  Number of sexual partners in the last year
Total number of sexual partners | up to 4 months
  Total number of sexual partners in the participants lifetime
Use of condoms and contraceptives | up to 4 months
  Frequency of usage of condoms and contraceptive methods
STDs screening | up to 4 months
  Frequency of STDs screening
STD testing centers | up to 4 months
  Knowledge of the location of STD testing centers
Exclusive or non-exclusive sexual relationships | up to 4 months
  Frequency of exclusive and non-exclusive sexual relationships

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Mexicano del Seguro Social, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data available.

REFERENCES:
- [Background] Aburto-Arciniega MB, Escamilla-Santiago RA, Diaz-Olavarrieta CA, Fajardo-Dolci GE, Urrutia-Aguilar ME, Arce-Cedeno A, Mota-Sanchez AA, Guevara-Guzman R. Sexual health educational intervention in medical students. Gac Med Mex. 2020;156(2):164-170. doi: 10.24875/GMM.M20000354. PMID 32285861
- [Background] Campero Cuenca L, Atienzo EE, Suarez Lopez L, Hernandez Prado B, Villalobos Hernandez A. [Sexual and reproductive health among adolescents in Mexico: evidence and proposals]. Gac Med Mex. 2013 May-Jun;149(3):299-307. No abstract available. Spanish. PMID 23807332
- [Background] Cuffe KM, Newton-Levinson A, Gift TL, McFarlane M, Leichliter JS. Sexually Transmitted Infection Testing Among Adolescents and Young Adults in the United States. J Adolesc Health. 2016 May;58(5):512-9. doi: 10.1016/j.jadohealth.2016.01.002. Epub 2016 Mar 15. PMID 26987687
- [Background] Cifuentes E, Trasande L, Ramirez M, Landrigan PJ. A qualitative analysis of environmental policy and children's health in Mexico. Environ Health. 2010 Mar 23;9:14. doi: 10.1186/1476-069X-9-14. PMID 20331868
- [Background] Goyal MK, Teach SJ, Badolato GM, Trent M, Chamberlain JM. Universal Screening for Sexually Transmitted Infections among Asymptomatic Adolescents in an Urban Emergency Department: High Acceptance but Low Prevalence of Infection. J Pediatr. 2016 Apr;171:128-32. doi: 10.1016/j.jpeds.2016.01.019. Epub 2016 Feb 2. PMID 26846572
- [Background] Friedman AL, Kachur RE, Noar SM, McFarlane M. Health Communication and Social Marketing Campaigns for Sexually Transmitted Disease Prevention and Control: What Is the Evidence of their Effectiveness? Sex Transm Dis. 2016 Feb;43(2 Suppl 1):S83-101. doi: 10.1097/OLQ.0000000000000286. PMID 26779691
- [Background] Uken RB, Brummer O, von Schubert-Bayer C, Brodegger T, Teudt IU. Oral HPV prevalence in women positive for cervical HPV infection and their sexual partners: a German screening study. Eur Arch Otorhinolaryngol. 2016 Jul;273(7):1933-42. doi: 10.1007/s00405-016-3953-1. Epub 2016 Mar 9. PMID 26961518
- [Background] Mohammed H, Mitchell H, Sile B, Duffell S, Nardone A, Hughes G. Increase in Sexually Transmitted Infections among Men Who Have Sex with Men, England, 2014. Emerg Infect Dis. 2016 Jan;22(1):88-91. doi: 10.3201/eid2201.151331. PMID 26689861
- [Background] Pearson WS, Peterman TA, Gift TL. An increase in sexually transmitted infections seen in US emergency departments. Prev Med. 2017 Jul;100:143-144. doi: 10.1016/j.ypmed.2017.04.028. Epub 2017 Apr 26. PMID 28455221